CLINICAL TRIAL: NCT01684085
Title: Explanation About Sleep Given After Traumatic Event, and Its Effect on the Trajectory of Post Traumatic Stress Disorder (PTSD)
Brief Title: Explanation About Sleep in Post Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHEBA-12-9175-JZ-CTIL
Record Dates: First submitted 2012-09-05; First posted 2012-09-12 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Post Traumatic Stress Disorder; Sleep Deprivation
Keywords: sleep deprivation, PTSD,prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Deprivation | interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Encouragement to sleep (Placebo Comparator): Encouraging explanation to sleep, rest and receiving Lorazepam 1mg in the first night post trauma
  Interventions: Behavioral: Explanation encouraging sleep; Drug: Lorazepam
- Encouragement to deprived sleep (Experimental): Encouraging explanation to deprived sleep in the first night post trauma
  Interventions: Behavioral: Explanation discouraging sleep

INTERVENTIONS:
Behavioral: Explanation encouraging sleep — An explanation will be given about sleep, encouraging the patient to sleep - lorazepam 1mg will be offered to promote sleep.
  Arms: Encouragement to sleep
Behavioral: Explanation discouraging sleep — An explanation about sleep will be given, discouraging the patient from sleeping in the first night after the traumatic event.
  Arms: Encouragement to deprived sleep
Drug: Lorazepam — Lorazepam 1 mg
  Arms: Encouragement to sleep

SUMMARY:
This study is designed to test the effect of an explanation about the first sleep following trauma exposure, on the development of Post Traumatic Stress Disorder (PTSD) in the months following the traumatic event.

DETAILED DESCRIPTION:
This is a Single blind, prospective, placebo controlled trial in which trauma victims are randomized to receive an explanation about the first sleep following trauma exposure.

To provide a baseline prior the explanation, participants will receive a medical and psychological evaluation. at this point the participants will be given one of two explanations about sleep. The experimental group will receive an encouragement to deprived sleep explanation, and the control group will receive an encouragement to sleep explanation, Lorazepam 1mg will be offered to assist sleep. After two weeks the research assistant or study psychiatrist will perform behavioral ratings and complete history details pertaining to PTSD risk factors. Participants will be assessed again by the study psychiatrist or research assistants at 1 & 3 months. Further assessments might be done at 6 & 13 months.

Eligible subjects will include men and women age 18-70, who have been exposed to an event meeting the DSM-IV "A.1" criterion for trauma exposure, and who provide written, informed consent to participate in the study.

Potential participants will be recruited from trauma victims who arrived at the Chaim Sheba Medical Center Emergency Room.

ELIGIBILITY:
Inclusion Criteria:

1. Persons age 18-70, who have been exposed to an event meeting the DSM-IV "A.1" criterion for trauma exposure.
2. Persons who arrived at the Chaim Sheba Medical Center Emergency Room.
3. Who provide written, informed consent to participate in the study -

Exclusion Criteria:

1. Physical injury that would contraindicate participation or interfere with a subject's ability to give informed consent or cooperate with the screening or collection of initial measures. Examples include severe burn injury, life-threatening medical or surgical condition, condition requiring surgical intervention under general anesthesia, as indicated by clinical judgment;
2. Traumatic exposure that reflects ongoing victimization (e.g., domestic violence) to which the subject is likely to be re-exposed during the study period.
3. Overt psychopathology, intoxication, or under the influence of substances.
4. Evidence or history of schizophrenia, bipolar, other psychotic condition;
5. Prior history of PTSD;
6. Current or past history of dementia, amnesia, or other cognitive disorder predating trauma exposure;
7. Assessed serious suicide risk. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
PTSD severity as measured by CAPS | 4 months
  The primary outcome is PTSD severity at the end of the trial .This will be determined using the Clinician Administered PTSD Scale (CAPS), a scale with established reliability and good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Department of Psychiatry, Chaim Sheba Medical Center, Israel
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel